CLINICAL TRIAL: NCT03763968
Title: Multicentre REtrospective StuDy of Treatment and OUtComes in ST-elevatION Myocardial Infarction(STEMI) Patients in Fujian Province
Brief Title: Multicentre REtrospective StuDy of Treatment and OUtComes in STEMI Patients in Fujian Province
Acronym: REDUCTION
Status: Completed | Type: Observational
Sponsor: Yan-song Guo (Other)
Collaborators: Longyan City First Hospital (Other); The Affiliated Hospital of Putian University (Other); The Second Affiliated Hospital of Fujian Medical University (Other); The MinDong Hospital of Ningde City (Unknown)
Responsible Party: Sponsor-Investigator, Yan-song Guo, Fujian Provincial Hospital, Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Other Study IDs: YGuo
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Treatment Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: treatment and outcome

SUMMARY:
This is a multicentre observational study planned to gather follow up data for a period of 1 year in order to understand the treatments and outcomes of ST-segment elevation myocardial infarction(STEMI) and improve medical care quality in Fujian province for China. Consecutive patients who were admitted and diagnosed with STEMI between January 2014 December 2018 were conducted at five regional representative hospitals in Fujian province, which included the Fujian Provincial Hospital,Longyan First Hospital, the affiliated hospital of putian university,the Second Affiliated Hospital of Fujian Medical University and Mindong Hospital of Ningde City.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients with symptom onset within 30 days

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: STEMI patients with symptom onset within 30 days
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 5years
  all mortality,cardiovascular mortality

SECONDARY OUTCOMES:
other in-hospital complications | 5years
  recurrent myocardial infarction, target vessel revascularization,contrast-induced acute kidney injury,stroke,bleeding,and so on
MACEs for long-term follow up | 1 year
  mortality,stent restenosis, recurrent myocardial infarction, and target vessel revascularization,stroke,bleeding,and so on

CONTACTS AND LOCATIONS:
Overall Officials: Kai-yang Lin, Doctor, Principal Investigator — Fujian Provincial Hospital
Locations (1):
- Fujian Provincial, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No